CLINICAL TRIAL: NCT00393835
Title: A Multicenter, Non-Randomized, Open Label Trial Of Azithromycin Sustained Release (SR) For The Treatment Of Laryngopharyngitis or Tonsillitis or Acute Bacterial Rhinosinusitis In Japan Adults
Brief Title: A Trial Of Azithromycin SR For The Treatment Of Laryngopharyngitis or Tonsillitis or Acute Bacterial Rhinosinusitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0661176
Record Dates: First submitted 2006-10-26; First posted 2006-10-30 (Estimated); Last update posted 2008-05-16 (Estimated); Status verified 2008-05

CONDITIONS: Upper Respiratory Tract Infection
MeSH Terms: conditions — Respiratory Tract Infections

INTERVENTIONS:
Drug: Azithromycin SR

SUMMARY:
To evaluate the clinical efficacy and safety in patients with Laryngopharyngitis or Tonsillitis or Acute Bacterial Rhinosinusitis receiving a dose of 2 g of azithromycin in the SR formulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed Laryngopharyngitis or Tonsillitis or Acute Bacterial Rhinosinusitis

Exclusion Criteria:

* Severe underlying disease; patients in which drug clinical evaluation is difficult because of confounding diseases.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2006-11; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is Investigator's Clinical efficacy at Day 8.

SECONDARY OUTCOMES:
Endpoints of efficacy are as follows: Investigator's clinical efficacy (at Day 4, Day 15 and 29) Bacteriological efficacy (at Day 4, 8, 15 and 29) Safety Endpoints: Adverse events and safety Laboratory data

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Japan (4):
  - Pfizer Investigational Site, Gobō, Wakayama
  - Pfizer Investigational Site, Hashimoto, Wakayama
  - Pfizer Investigational Site, Shinjo-cho, Tanabe, Wakayama
  - Pfizer Investigational Site, Wakayama, Wakayama

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661176&StudyName=A%20Trial%20Of%20Azithromycin%20SR%20For%20The%20Treatment%20Of%20Laryngopharyngitis%20or%20Tonsillitis%20or%20Acute%20Bacterial%20Rhinosinusitis